CLINICAL TRIAL: NCT00222625
Title: Randomized, Open, Prospective, Multicenter Pilot Study to Evaluate the Efficacy and Safety of Activated Recombinant Factor VII in Acute Intracerebral Haemorrhage in Patients Treated With Oral Anticoagulants or Antiplatelets Agents.
Brief Title: rFVIIa in ICH in Patients Treated With Anticoagulants or Anti-Platelets
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-002155-40; 04 MICV AI 04
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Oral Anticoagulants; Antiplatelet Agents; Recombinant Activated Factor VII
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — recombinant FVIIa

INTERVENTIONS:
Drug: rFVIIa + (vit K in AO patients)
Drug: FFP or aPCC+ vit K in AO treated patients

SUMMARY:
Evaluation of efficacy and safety of recombinant factor VIIa versus standard therapy in preventing early haematoma growth in spontaneous acute intracerebral haemorrhage in patients treated with oral anticoagulants or antiplatelets agents

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is the deadliest, most disabling, and least treatable form of stroke. Approximately 40% of patients die within 1 month of ICH onset, and two-thirds of survivors never regain functional independence. Though guidelines for supportive care exist, there is currently no treatment that has been shown in a randomized-controlled trial to definitely improve outcome after ICH. Hematoma volume is a critical determinant of mortality and functional outcome after ICH, and early hematoma growth may be an important cause of early neurological deterioration.

Considerable clinical interest has been given to the relationship between antiplatelet and antithrombotic treatment and ICH.

The reported incidence of major bleeding events in patients undergoing antithrombotic treatment is 5-11/1,000 patients/year, while the overall range of hemorrhages is about 62/1,000 patients/year.In the patients treated with antithrombotic drugs (oral anticoagulants or antiplatelets agent) the incidence rate of ICH has been shown higher than in the general population. Moreover, the mortality rate for both spontaneous and post-traumatic events is higher in antithrombotic treated patients than in controls. [14,15] rFVIIa has been successfully used to control ICH in patients with hemophilia or other coagulation disorders, and can arrest intraoperative bleeding and reverse coagulopathies in patients undergoing neurosurgical procedures.[19] rFVIIa has also been reported to prevent or minimize refractory bleeding in non-coagulopathic patients.

ELIGIBILITY:
Inclusion Criteria:

* ICH in patient on treatment with one of the following:
* a)oral anticoagulant (INR upper than 1,4 at enrollment
* b) aspirin, whatever dosage
* Male or female subjects, age > 18 years.
* Informed consent

Exclusion Criteria:

* INR below 1.4 for patients on oral anticoagulants.
* Patients with secondary ICH related to infarction, tumor, cerebrovenous thrombosis, thrombolysis.
* Planned neurosurgical intervention.
* Any history of haemophilia or other congenital or acquired coagulopathy requiring specific antihemorrhagic treatment.
* Acute myocardial ischaemia or acute thrombotic stroke (within one year).
* Septicemia, intravascular disseminated coagulation.
* Pregnancy.
* Limb amputation due to vascular disease or claudication within last 30 days.
* Known or suspected allergy to the trial product or related products.
* Participation in other trials within the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2005-09; Study Completion 2006-09

PRIMARY OUTCOMES:
EFFICACY: change in ICH volume from prior to dosing to 24 hours
SAFETY: occurrence of clinical adverse events (Thromboembolic events, death)

SECONDARY OUTCOMES:
Difference between groups on the modified Rankin Scale, the Barthel Index (BI), the Extended Glasgow Scale (EGCS), and the National Institute of Health's Stroke Scale (NIHSS) at one and three month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Iorio, Principal Investigator — University Of Perugia
Locations (9):
- Italy (9):
  - A.O.R.N. San Sebastiano, Caserta
  - Emergency Room, Forlì
  - Emergency Department - S.Martino Hospital, Genoa
  - Emergency Room - University of Messina, Messina
  - Internal and Vascular Medicine - Stroke Unit - University of Perugia, Perugia
  - Divisione di Neurologia, Piacenza
  - Emergency Room, Ravenna
  - Emergency Room, Reggio Emilia
  - Stroke Unit - Policlinico Universitario Umberto I, Rome

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Iorio A. Iatrogenic causes of an ICH: OAT therapy. Eur J Anaesthesiol Suppl. 2008;42:8-11. doi: 10.1017/S0265021507003171. PMID 18289410